CLINICAL TRIAL: NCT06249282
Title: A Phase I Clinical Trial of Carfilzomib in Combination With Sotorasib in Patients With KRASG12C Mutated Advanced Non-Small Cell Lung Cancer
Brief Title: Carfilzomib in Combination With Sotorasib for the Treatment of Patients With KRAS G12C Mutated Advanced or Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23477; NCI-2023-11093 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23477 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-01-11; First posted 2024-02-08 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Biopsy; Specimen Handling; carfilzomib; Magnetic Resonance Spectroscopy; sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (carfilzomib, sotorasib) (Experimental): Patients receive carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16 of each cycle and sotorasib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO at screening and undergo CT or MRI and collection of blood samples at screening and on study. Patients may undergo optional biopsies on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Carfilzomib; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Magnetic Resonance Imaging; Drug: Sotorasib

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carfilzomib — Given IV
  Other Names: Carfilnat; CFZ; Kyprolis; PR-171
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Sotorasib — Given PO
  Other Names: AMG 510; AMG-510; AMG510; Lumakras; Lumykras

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of carfilzomib in combination with sotorasib in treating patients with KRAS G12C-mutated non-small cell lung cancer (NSCLC) that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). Carfilzomib is a drug that binds to and inhibits the activity of the protein complex that is responsible for degrading other damaged or unneeded proteins. The inhibition of this protein by carfilzomib can then cause tumor growth inhibition and cell death. Sotorasib is a drug that binds to and inhibits the activity of the KRAS G12C mutant. This may inhibit growth in KRAS G12C-expressing tumor cells. Combining carfilzomib and sotorasib may be a safe and effective treatment option for patients with KRAS G12C-mutated advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of the combination of carfilzomib and sotorasib in KRAS G12C mutated NSCLC following progression on KRAS inhibitor.

II. Describe the safety of the combination of carfilzomib and sotorasib in KRAS G12C mutated NSCLC following progression on KRAS inhibitor.

SECONDARY OBJECTIVES:

I. Describe clinical responses at all dose levels, including the recommended dose level using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.

II. Describe other efficacy endpoints, including progression-free survival (PFS), duration of response (DOR), and overall survival (OS) at the recommended dose level.

EXPLORATORY OBJECTIVES:

I. Evaluate the pharmacokinetics of the combination of carfilzomib and sotorasib.

II. Explore biomarkers of response and resistance through tumor biopsies and circulating tumor deoxyribonucleic acid (ctDNA).

OUTLINE: This is a dose-escalation study of carfilzomib in combination with (fixed-dose) sotorasib.

Patients receive carfilzomib intravenously (IV) over 30 minutes on days 1, 2, 8, 9, 15, and 16 of each cycle and sotorasib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) at screening and undergo computed tomography (CT) or magnetic resonance imaging (MRI) and collection of blood samples at screening and on study. Patients may undergo optional biopsies on study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed NSCLC that is metastatic or advanced. The tumor must exhibit evidence of KRASG12C mutation which is determined by either a Clinical Laboratory Improvement Act (CLIA) certified ctDNA assay or by a CLIA certified tumor tissue assay
* Measurable disease by RECIST v1.1
* Failed prior KRAS inhibitor
* Fully recovered from the acute toxic effects (except alopecia) from prior anti-cancer therapy
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate central nervous system (CNS) specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3 (performed within 14 days prior to day 1 of protocol therapy)

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Hemoglobin (Hb) ≥ 9 g/dL (performed within 14 days prior to day 1 of protocol therapy)
* Platelets ≥ 100,000/mm^3 (performed within 14 days prior to day 1 of protocol therapy)

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease) (performed within 14 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) ≤ 3 x ULN (or ≤ 5 x ULN in the setting of liver metastatic disease) (performed within 14 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) ≤ 5 x ULN (or ≤ 5 x ULN in the setting of liver metastatic disease) (performed within 14 days prior to day 1 of protocol therapy)
* Creatinine clearance of ≤ 1.5 x ULN or glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2 (performed within 14 days prior to day 1 of protocol therapy)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (performed within 14 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 120 days after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Chemotherapy or immunotherapy within 21 days prior to day 1 of protocol therapy
* Radiation therapy within 14 days prior to day 1 of protocol therapy
* KRAS inhibitor within 14 days prior to day 1 of protocol therapy
* Investigational therapy within 28 days prior to day 1 of protocol therapy (or 5 half-lives, use whichever is shorter)
* Inability to previously tolerate (240 mg, QD) sotorasib
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Clinically significant uncontrolled illness
* Evidence of chronic hepatitis B virus (HBV) infection and HBV viral load detectable
* Evidence of untreated chronic hepatitis C virus (HCV) infection. Patients with HCV infection currently on treatment are eligible if they have an undetectable HCV viral load
* Active infection requiring antibiotics (not to be completed by day 1 of protocol therapy)
* Known history of immunodeficiency virus (HIV) with detectable viral load
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* New York Heart Association (NYHA) class III or IV heart failure, myocardial infarction in the preceding 6 months, conduction abnormalities uncontrolled by medications
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | During cycle 1 (each cycle is 28 days)
  The incidence of dose-limiting toxicities during cycle 1 will be used to determine the maximum tolerated dose and the recommended phase II dose of the comibination of carfilzomib and sotorasib. Will be described and graded at all dose levels using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Incidence of grade 3 and 4 treatment-related toxicities | Up to 30 days after completion of study treatment
  Grade 3 and 4 adverse events will be described and graded at all dose levels using the NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Objective response rate | From the start of treatment until disease progression/recurrence, assessed up to 30 days after completion of study treatment
  Defined as the proportion of all subjects with confirmed partial response or complete response, according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Response rate will be summarized by frequencies and percentages, along with the corresponding exact 95% confidence intervals.
Duration of response | From treatment response to progression or death, assessed up to 30 days after completion of study treatment
  Will be estimated using the Kaplan-Meier method.
Progression-free survival | From day 1 of treatment until the criteria for disease progression is met or until death, assessed up to 30 days after completion of study treatment
  Disease progression will be defined using RECIST version 1.1. Will be estimated using the Kaplan-Meier method.
Overall survival | From the date of study enrollment to the date of death, assessed up to 30 days after completion of study treatment
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Salgia, MD, Principal Investigator — City of Hope Medical Center; Jyoti Malhotra, MD (Co-PI), Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California